CLINICAL TRIAL: NCT06845878
Title: A Conversational Agent to Support Follow-up Care for Individuals in Recovery for Substance Use Disorder
Brief Title: A Chatbot to Support Substance Use Recovery
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dimagi Inc. (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); University of California, Los Angeles (Other); Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2R44DA050218 (NIH); 2R44DA050218-02 (NIH)
Record Dates: First submitted 2025-02-18; First posted 2025-02-25 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-02

CONDITIONS: Opiate-Related Disorders; Opiate Substitution Treatment

STUDY DESIGN:
Intervention Model Description: Pre-Post Intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Chatbot (Experimental): Participants will receive access to a chatbot for 12 weeks that can be used from a mobile device to support follow-up care and recovery needs.
  Interventions: Other: chatbot

INTERVENTIONS:
Other: chatbot — Participants will:
  * Participate in a baseline session to complete an initial survey and get trained on using the chatbot
  * Use the chatbot for 12 weeks and submit a brief weekly survey to provide feedback
  * Complete a final survey to provide substance use and health information as well as give feedback on the experience using the chatbot
  * Allow access to a limited set of demographic, substance use and health information in electronic health record for study analyses and context.
  Other Names: Suzy; conversational agent

SUMMARY:
The goal of this clinical trial is to learn if/how an AI chatbot can support patients who in recovery for substance use, specifically those who are receiving medication for opioid use disorder.

Can the chatbot help lower drug use? Can the chatbot help improve clinical appointment adherence? Can the chatbot help patients build self-efficacy in leading their own recovery journey? Will the chatbot help reduce workload burden for primary care teams? Can the chatbot serve as a safe, useful and engaging tool to support patients?

Researchers will investigate the effects of using a chatbot to support follow-up care for patients in opioid use recovery.

Participants will:

* Receive access to a chatbot for 12 weeks that they can use to prepare for upcoming clinical appointments, find community resources, learn about urge-surfing and wellness techniques, and query for assistance with other recovery-related information and tasks
* Complete surveys and provide user feedback

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Comfortable with reading, understanding, and communicating in English
* Receiving medication treatment for OUD at MGH?
* Able to participate in a remote interview?
* Own or have reliable access to Wi-Fi or a cellular network
* Willing to use a mobile device to access the chatbot?

Exclusion Criteria:

* Has any cognitive, visual, or auditory impairments that may prevent the participant from using the chatbot on a mobile device?
* Unstable medical condition that compromises the ability to safely participate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2025-03-07 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Change in SUD severity | 12 weeks
  Addiction Severity Index (ASI) Drugs composite score; Scored 0-7 with higher scores indicating increasing severity
Change in psychological health (Anxiety) | 12 weeks
  General Anxiety Disorder-7 (GAD-7); scored 0-21 with higher scores indicating increasing anxiety
Change in psychological health (Depression) | 12 weeks
  Patient Health Questionnaire-8 (PHQ-8); scored 0-24 with higher scores indicating more severe depression
Change in self-efficacy for managing chronic conditions (Emotions) | 12 weeks
  PROMIS Short Form 8a (Managing Emotions); scored from 8-40 with higher scores indicating higher confidence managing emotions
Change in self-efficacy for managing chronic conditions (Social Interactions) | 12 weeks
  PROMIS Short Form 8a (Social Interactions); scored from 8-40 with higher scores indicating higher confidence with managing social interactions

SECONDARY OUTCOMES:
Change in quality of life | 12 weeks
  World Health Organization Quality of Life (WHOQoL-BREF) Assessment; higher scores indicate higher quality of life
Change in social needs | 12 weeks
  Accountable Health Communities Health-Related Social Needs (AHC HRSN) screening; higher scores indicate higher unmet social needs
Chatbot usability | End of 12 week intervention
  Chatbot Usability Questionnaire (CUQ); scored 0-100 with higher scores indicating higher usability
User Satisfaction | End of 12 week intervention
  Net Promoter Score (NPS); scored -100 to 100 with higher scores indicating higher user satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Y. Xian Ho, PhD, Principal Investigator — Dimagi Inc.; Jonathan Jackson, MEng, Principal Investigator — Dimagi Inc.
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
This study will include sensitive data from a small sample of patients with experience with substance use therefore data will be reported in aggregate and only qualitative data collected from participants may be reported individually and anonymously.